CLINICAL TRIAL: NCT05375721
Title: ST36 Acupoint Injection With Anisodamine for Postoperative Nausea and Vomiting in Women Following Bariatric Surgery: A Multicentre, Randomised, Double-Blind Controlled Trial.
Brief Title: Prevention of PONV With Traditional Chinese Medicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Anhui Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Huashan Hospital (Other); Henan Provincial People's Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); First Affiliated Hospital of Jinan University (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, hui hou, Principal Investigator, The Second Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YX2021-152（F1）
Record Dates: First submitted 2022-04-22; First posted 2022-05-17 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: postoperative nausea and vomiting; bariatric surgery; Zusanli; anisodamine; obesity
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ST36 acupoint injection group (Experimental): Patients in this group will received bilateral ST36 injection with scopolamine 1ml/point
  Interventions: Procedure: ST36 acupoint injection
- pharmacoprophylaxis group (Placebo Comparator): Patients in this group will received bilateral ST36 acupoint injection with normal saline 1ml/point
  Interventions: Procedure: ST36 acupoint injection

INTERVENTIONS:
Procedure: ST36 acupoint injection — ST36 is located on the lateral surface of leg, 3 cun distal to the lower border of the patella, 1 finger-breadth lateral to the anterior crest of the tibia, between the tibialis anterior muscle and the tendon of the extensor digitorum longus. (The breadth of patient's middle finger was the proportional unit of measure "the cun", defined as the distance between the two medial ends of the creases of the interphalangeal joints when the patient's middle finger is flexed).

SUMMARY:
Postoperative nausea and vomiting (PONV) is particularly one of the most common complications after laparoscopic sleeve gastrectomy (LSG). It can lead to serious adverse events and delayed activity, and prolong the time of rehabilitation and discharge. Numbers of studies have been focused on identifying risk factors and therapies of PONV. Unfortunately, there' no consistent comments for PONV prevention in women after LSG. Notably, Zusanli (ST36) acupoint and anisodamine have been evidenced to treat various gastrointestinal conditions. The primary outcome of this study was to evaluate the impact of anisodamine injection in ST36 on PONV in women following bariatric surgery.

DETAILED DESCRIPTION:
At the onset of this investigation, we have already identified several methodologic issues, such as the timing of the acupuncture intervention, sample size, perioperative anesthetic techniques, and appropriate control groups. All subjects were randomly assigned to the following two groups: ST36 acupoint injection group (bilateral ST36 acupoint injection with scopolamine); pharmacoprophylaxis group (bilateral ST36 injection with normal saline). The primary outcome of this study was the total incidence of PONV during the hospital and after the discharge. Participants were randomly assigned into different groups according to the computer-generated randomization sequence (http://www.randomization.com). Patients, surgeons, care givers, anesthesiologists, nursing staff, and outcomes assessor, were all blinded to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with an American Society of Anesthesia (ASA) physical status I-IV
2. Scheduled for elective bariatric surgery
3. Written informed consent was obtained

Exclusion Criteria:

1. Patients with contraindications for acupoint injection
2. Difficulty in communicating with patients
3. Allergic diathesis for drugs used in the study or serious illness (heart, lung, kidney, or liver, et. al)
4. Coagulation dysfunction
5. Pre-existing psychological or neurological disorder
6. Pre-use medicine before surgery that would interferenced objective assessment (including the use of opioids, antiemetics or glucocorticoids)
7. Gastroesophageal reflux disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of PONV | At 0-2 hours after surgery
  The incidence and severity of PONV after bariatric surgery
The incidence and severity of PONV | At 2-6 hours after surgery
  Total usage of rescue antiemetic drugs after bariatric surgery
The incidence and severity of PONV | At 6-12 hours after surgery
  The incidence and severity of PONV after bariatric surgery
The incidence and severity of PONV | At 12-24 hours after surgery
  The incidence and severity of PONV after bariatric surgery
The usage of rescue antiemetic drugs | During 3 months after bariatric surgery
  Total usage of rescue antiemetic drugs after bariatric surgery

SECONDARY OUTCOMES:
15-item Quality of Recovery(QoR-15) | Postoperative 24 hours
  QoR-15 will be used to evaluate recovery quality after anesthesia, including 15 items covering sleep, satisfaction, emotion and pain et. al,total score ranges from 0 to 150,the higher score means the higher quality of recovery.
Postoperative pain | At 0-24 and 24-72 hours after surgery
  Patients will be asked about their pain level at rest and moving on a numeric rating scale (0=no pain,10=worst pain imaginable) .
Consumption of analgesics | During 3 months after bariatric surgery
  Cumulative analgesic consumption after surgery
Ambulation time | Postoperative 1-3 days
  Interval time of patients' transit from bed rest to ambulation after surgery
Postoperative food and water intake time | Postoperative 1-3 days
  Duration of eating and drinking after surgery
Postoperative hospitalization duration | 2 weeks after surgery
  Days of hospital staying after surgery
Pittsburgh sleep quality index | Before surgery and at postoperative 3 months
  Pittsburgh sleep quality index will be used to evaluate quality of sleep. The higher score means the lower quality of sleep.
Gastrointestinal Symptom Rating Scale | Before surgery and at postoperative 3 months
  Gastrointestinal symptom rating scale (GSRS) will be used to assess gastrointestinal function. The score ranges from 0 to 45. The higher score means poorer gastrointestinal function .
Hamilton depression rating scale | Before surgery and at postoperative 3 months
  Hamilton depression scale (HAMD) will be used to assess depression. HAMD 24 item version score range 0-96. The higher score means the higher possibility of depression.
Hamilton anxiety rating scale | Before surgery and at postoperative 3 months
  Hamilton anxiety scale (HAM-A) will be used to assess anxiety. Total score ranges from 0 to 56, the higher the score is, the more serious the anxiety is.
The MOS item short from health survey ,SF-36 | Before surgery and at the postoperative 3 months.The scale consists of 36 items，divided into 8 sections，score of each section ranges from 0 to 100, the higher the score is, the healthier is.
  Concise health status scale

OTHER OUTCOMES:
Consumption of propofol | During the bariatric surgery
  The total consumption of propofol during the surgery
Consumption of remifentanil | During the surgery
  The total consumption of remifentanil during the surgery
Consumption of sufentanil | During the surgery and postoperative 1-3 days
  The total consumption of sufentanil during the surgery
Duration of anesthesia | At the end of anesthesia
  From beginning to the end of anesthesia
Duration of surgery | At the end of surgery
  From beginning to the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ye Zhang, M.D, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (7):
- China (7):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Huashan Hospital Affiliated to Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication are to be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will become available when summary data are published.
Access Criteria: ChunXia Huang and Ye Zhang will review requests and criteria to share IPD. Requests are to be sent by email to huangchunxia@ahmu.edu.cn or zhangye_hassan@sina.com.